CLINICAL TRIAL: NCT02635334
Title: Asthma in the Elderly: A Randomized, Double-Blind, Placebo-Controlled, Cross-Over Study of the Effect of Montelukast
Brief Title: Asthma in the Elderly: The Effect of Montelukast
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Rohr and Columbo Asthma, Allergy and Immunology Specialists, P.C. (Other)
Responsible Party: Principal Investigator, Michele Columbo, M.D., Principal Investigator, Rohr and Columbo Asthma, Allergy and Immunology Specialists, P.C.
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: SSRF2015-01
Record Dates: First submitted 2015-12-10; First posted 2015-12-18 (Estimated); Last update posted 2016-10-05 (Estimated); Status verified 2016-10

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — montelukast

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Montelukast 10 mg daily for 8 weeks (Experimental): Study subjects will take montelukast 10 mg orally daily for 8 weeks
  Interventions: Drug: Montelukast 10 mg orally; Other: Placebo
- Placebo daily for 8 weeks (Placebo Comparator): Study subjects will take placebo orally daily for 8 weeks
  Interventions: Drug: Montelukast 10 mg orally; Other: Placebo

INTERVENTIONS:
Drug: Montelukast 10 mg orally
  Other Names: Singulair
Other: Placebo

SUMMARY:
This is a pilot study of the effect of montelukast in subjects with asthma who are 65 years old and older. Montelukast is a leukotriene receptor antagonist U.S. F.D.A. approved for the treatment of asthma in subjects who are 12 month old and older. This study is being done because there has been no placebo controlled study of montelukast focused on this group of patients. Elderly asthmatics have been mostly ignored in asthma studies. They are more likely to be underdiagnosed, undertreated, and hospitalized for asthma when compared to younger asthmatics. The pathophysiology of asthma in the elderly is typically different than in younger patients. This is a double-blind, placebo-controlled, crossover study. Investigators plan to enroll thirty subjects who have been diagnosed with asthma for at least one year, are non smoker, and did not smoke for more than 10 pack/year of tobacco products in their lifetime. After a run-in period of one week, the study subjects will take montelukast 10 mg orally for 8 weeks first and then placebo for 8 weeks, or vice versa. Primary objectives of this study are to evaluate the effect of montelukast on asthma symptoms assessed by daily symptom scores, the Asthma Control Test and the number of puffs of albuterol, and spirometric values (FEV1). Secondary objectives include studying whether montelukast affects peripheral blood eosinophils counts and serum IgE levels.

ELIGIBILITY:
Inclusion Criteria:

* Asthma diagnosed for at least one year;
* Able to swallow small capsules.

Exclusion Criteria:

* Tobacco smoking for more than 10/pack years;
* Previous adverse reaction to montelukast or other leukotriene inhibitor;
* History of hypereosinophilic disorder other than atopic disease;
* Treatment with montelukast within 4 weeks from randomization;
* Asthma exacerbation or treatment with prednisone/other systemic steroid within 4 weeks from randomization.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 26 (Actual)
Dates: Start 2015-11; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Effect of montelukast on asthma symptoms assessed by daily symptom scores. | 8 weeks
Effect of montelukast on the Asthma Control Test. | 8 weeks
Effect of montelukast on number of puffs of albuterol used to relieve asthma symptoms. | 8 weeks
Effect of montelukast on lung capacity assessed by spirometry (FEV1). | 8 weeks

SECONDARY OUTCOMES:
Effect of montelukast on peripheral blood eosinophils counts. | 8 weeks
Effect of montelukast on total serum IgE. | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Michele Columbo, M.D., Principal Investigator — Rohr and Columbo Asthma, Allergy, and Immunology Specialists
Locations (1):
- Rohr and Columbo Asthma, Allergy and Immunology Specialists, P.C., Bryn Mawr, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No